CLINICAL TRIAL: NCT05269654
Title: A Single Center, Double-Blinded, Split-Body, Randomized Clinical Trial of Injectable Poly-L-Lactic Acid for Volumization and Adipogenesis of the Hip Dell
Brief Title: Injectable Poly-L-Lactic Acid for Volumization and Adipogenesis of the Hip Dell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Sherif Mikhail, MD, Research Director, Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sculptra Aesthetic - Hip Dell
Record Dates: First submitted 2022-02-04; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Skin Laxity
Keywords: Skin; Volume; Volume Loss; Hips; Cosmetic
MeSH Terms: conditions — Cutis Laxa | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-site, double-blinded, split-body, randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject and Outcome Assessor will be unaware of which side of the subject is treated with the study device and which is treated with saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- injectable poly-L-lactic acid (Experimental): One side of the subject's hips will be treated with injectable poly-L-lactic acid (PLLA, Sculptra® Aesthetic; Galderma Laboratories; Fort Worth, TX).
  Interventions: Device: injectable poly-L-lactic acid
- Normal Saline (Sham Comparator): One side of the subject's hips will be treated with injectable normal saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Device: injectable poly-L-lactic acid — Injectable biostimulant for volume loss
  Other Names: PLLA; Sculptra; Sculptra Aesthetic; Galderma
  Arms: injectable poly-L-lactic acid
Other: Normal Saline — Sham Comparator
  Arms: Normal Saline

SUMMARY:
To assess the safety, efficacy and subject satisfaction associated with volumization of the hip dell with injectable poly-L-lactic acid (PLLA), or Sculptra® Aesthetic (Galderma Laboratories, Fort Worth, TX).

DETAILED DESCRIPTION:
The primary objectives of this clinical trial is to assess efficacy of adipose tissue generation (adipogenesis) and volumization following treatment of the hip dell with injectable poly-L-lactic acid (PLLA, Sculptra® Aesthetic; Galderma Laboratories; Fort Worth, TX).

Enrolled subjects will be randomized to two (2) treatment groups: "right hip dell treated" and "left hip dell treated". All subjects will receive three (3), single-sided injections of Sculptra® Aesthetic (Galderma Laboratories; Fort Worth, TX), performed one (1) month ± 7 days apart. Treatments will be provided to one side randomly assigned to either "right side" or "left side". The non-treatment side will receive bacteriostatic saline, injected in the same manner as Sculptra® Aesthetic. One (1) vial of Sculptra® Aesthetic, diluted to 8mL, will be used per treatment session.

Subjects satisfying all inclusion and no exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory digital photography with overhead lighting and VECTRA® (Canfield Scientific, Inc.; Parsippany, NJ) 3D volumetric body photography will be obtained of each subject's treatment area. In order to participate in the study, subjects must provide written informed consent to have their photographs used for research, publication, and/or commercial purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 30 to 60 years
* Subjects in good general health based on investigator's judgment and medical history
* Moderate to severe hip dell volume deficit as determined by the investigators
* Must be willing to give and sign an informed consent form and photographic release form
* Must have a stable body weight for at least six (6) months prior to study entry
* Must be willing to maintain usual sun exposure, diet, and exercise routines for the duration of the study
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.
* A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
* Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.
* Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

* Liposuction to bilateral hips, flanks, thighs, buttocks during the 12-month period prior to study treatment or any time during the course of the study
* Mesotherapy, dermal fillers, biostimulatory injectables, fat grafting, radiofrequency device treatments, microfocused ultrasound device treatments, laser and light-based device treatments, microneedling, cryolipolysis, high intensity focused electromagnetic energy device treatment, or surgery (i.e., lower body lift, buttocks augmentation, abdominoplasty, etc.) during the 12-month period before study treatment c) Any investigational treatment for a volume deficit of the bilateral hip dell areas during the 12-month period before the study treatment d) Massage therapy during the 3-month period before study treatment. e) Creams/cosmeceuticals and/or home therapies to promote plumping of the bilateral hip dell area during the four-week period before study treatment f) Subjects with scarring in the treatment areas g) History of thrombosis, post-thrombosis syndrome, or any vascular disorder of the bilateral lower extremities
* Any history of bleeding or coagulation disorders i) Subjects with tattoos or permanent implants in the treatment areas j) Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* History of keloid or hypertrophic scarring
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas
* Subjects who spray tanned or used sunless tanners in the treatment areas four (4) weeks prior to study treatment
* History of lidocaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Subjects who are on an immunosuppressant or have an autoimmune condition
* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subjects must self-report as female
Enrollment: 20 (Estimated)
Dates: Start 2022-03-04 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Histological Analysis | Baseline to three months post final treatment
  Comparison of measure of adipose tissue in biopsies taken from device and sham treated areas prior to baseline and at followup visits
Histological Analysis | Baseline to six months post final treatment
  Comparison of measure of adipose tissue in biopsies taken from device and sham treated areas prior to baseline and at followup visits
Volumetric Analysis | Pre-Treatment Visit 2/ Baseline
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Pre-Treatment Visit 3/ Day 14
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Pre-Treatment Visit 4/ Day 44
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Pre-Treatment Visit 5/ Day 74
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Visit 6/ Day 104
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Visit 7/ Day 164
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Visit 9/ Day 254
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Volumetric Analysis | Visit 11/ Day 344
  Analysis of tissue volume in treatment zones based on measurements obtained via 3D photography
Physician Global Aesthetic Improvement Scale | 1 Month Follow-Up visit
  Blinded-Evaluator assessment of change in appearance of treated areas where 1 + Very Much Improved, 2 = Much Improved, 3 = Improved, 4 = No Change, and 5 = Worse
Physician Global Aesthetic Improvement Scale | 3 Month Follow-Up visit
  Blinded-Evaluator assessment of change in appearance of treated areas where 1 + Very Much Improved, 2 = Much Improved, 3 = Improved, 4 = No Change, and 5 = Worse
Physician Global Aesthetic Improvement Scale | 6 Month Follow-Up visit
  Blinded-Evaluator assessment of change in appearance of treated areas where 1 + Very Much Improved, 2 = Much Improved, 3 = Improved, 4 = No Change, and 5 = Worse
Physician Global Aesthetic Improvement Scale | 9 Month Follow-Up visit
  Blinded-Evaluator assessment of change in appearance of treated areas where 1 + Very Much Improved, 2 = Much Improved, 3 = Improved, 4 = No Change, and 5 = Worse
Identification of correct Treatment Area (Right vs Left Hip) | 9 Month Follow-Up visit
  Blinded-Evaluator performed assessment of which side received study treatment and which received sham

SECONDARY OUTCOMES:
Collagen Analysis | Upon analysis of biopsies collected at Day 0 and 3 and 6 Month Follow-Up visits
  Quantitative analysis of collagen amounts based on histology
Elastin Analysis | Upon analysis of biopsies collected at Day 0 and 3 and 6 Month Follow-Up visits
  Quantitative analysis of elastin amounts based on histology
Skin Thickness | Day 0 and 3, 6, and 9 Month Follow-Up visits
  Ultrasound imaging measurements of skin thickness/thickness of dermis
Subject Global Aesthetic Improvement Score | 1, 3, 6, and 9 Month Follow-Up visits
  Subject assessment of change in appearance of treated areas rated numerically from 1 to 5 with 1 being very much improved to 5 being worse
Subject Satisfaction Questionairre | 1, 3, 6, and 9 Month Follow-Up visits
  Degree of subject satisfaction with treatment outcomes rated numerically from 0 to 4 with 0 being not satisfied to 4 being extremely satisfied
Evaluation of Side Effects | Day 44, Day 74, Day 104, Day 164, Day 178, Day 254, Day 268, Day 433
  Assessment of treatment related adverse events by Investigator

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center/Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided